CLINICAL TRIAL: NCT01438164
Title: Estudo de Custo-efetividade Para o Sistema único de Saúde - SUS Sobre o Exame de Metabolismo de Glicose Marcada Com Flúor-18 Pela Tomografia de emissão de pósitron-PET
Brief Title: Cost-effectiveness of FDG-PET
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Collaborators: Netherlands: Ministry of Health, Welfare and Sports (Other Government)
Responsible Party: Principal Investigator, Juliano Julio Cerci, Pesquisador executante, University of Sao Paulo
Other Study IDs: USP0460/05
Record Dates: First submitted 2011-09-20; First posted 2011-09-21 (Estimated); Last update posted 2011-09-21 (Estimated); Status verified 2011-09

CONDITIONS: Oncologic Patients
Keywords: FDG-PET; cancer; staging; Evaluate the cost impact in the evaluation of oncologic patients.
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- oncologic patients: initial staging

SUMMARY:
Evaluation of cost-effectiveness of FDG-PET for the public health system in Brazil.

DETAILED DESCRIPTION:
To provide detailed information about cost and effectiveness of FDG-PET in multiple oncological diseases, such as Lymphoma, lung cancer and esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Cancer

Exclusion Criteria:

* Other malignancy
* Uncontrolled Diabetes
* Pregnancy

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 500 oncologic patients
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2005-06; Primary Completion 2010-06 (Actual); Study Completion 2011-09 (Actual)